CLINICAL TRIAL: NCT05227950
Title: Usefulness of Cell-free DNA Quantification With Fluorescent Assay in Response Evaluation of Palliative Chemotherapy
Brief Title: Cell-free DNA Quantification for Predictive Marker of Palliative Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kwonoh Park, MD phD, Assistant professor, Pusan National University Yangsan Hospital
Other Study IDs: CFD-3
Record Dates: First submitted 2022-01-24; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Cell-Free Nucleic Acids; Biomarkers; Fluorescence; Palliative Chemotherapy
Keywords: cell-free nucleic acids; biomarkers; palliative chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — quantification of fluorescence based cell-free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is design to address, as follows:

1. correlation between fluorescence-based CFD measurements and tumor burden (primary tumor size, number of metastatic sites)
2. fluorescence-based CFD measurements and changes are related to tumor response. Based on the results of this study, the role of fluorescence-based CFD as a predictive biomarker for palliative chemotherapy is to be confirmed.

DETAILED DESCRIPTION:
* It is important to check the response to chemotherapy. Currently, it is mostly evaluated as a radiologic response or, rarely the change of tumor markers.
* In the case of radiologic response tests at intervals of 6-8 weeks, there are cases where the economic burden and radiation exposure risk, additionally evaluation lesion is lack in a few case. Except for prostate cancer and ovarian cancer, the majority of carcinomas do not have cancer markers for assessing treatment response. Therefore, there is a need for biomarkers that can predict the response of anticancer treatment.
* In many studies, it has been reported that various types of circulating cell free DNA (CFD) are increased in various cancer types.
* Recently, a fluorescence based CFD method that can directly measure nucleic acids without a DNA extraction process has been developed, which makes testing simpler and more economical, and can be conveniently applied to cancer diagnosis and treatment response.
* This study is plan to evaluate the relationship between fluorescence-based CFD and treatment response in patients starting palliative chemotherapy, and check whether it can serve as a response evaluation for palliative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed initially metastatic or recurrent cancer who are expected to undergo primary palliative chemotherapy (patients who relapse after adjuvant chemotherapy before/after existing surgery can also be enrolled regardless of period)
* Patients with definitive tumor burden (Patients who do not have residual lesions due to metastasectomy are excluded. However, measurable lesions according to RECIST 1.1 are not mandatory, and evaluable lesions are possible)
* ECOG PS 0-2
* Adequate bone marrow, renal function, liver function to receive chemotherapy
* Patients with informed consent form

Exclusion Criteria:

* Patients with treating antibiotic treatment within 3 days of study enrollment due to overt or suspected infection
* Other serious illness or medical condition

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed initially metastatic or recurrent cancer who are expected to undergo primary palliative chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
relationship between CFD and tumor burden | 2 year
  Confirmation of relationship between baseline CFD value and primary tumor size and number of metastatic sites

SECONDARY OUTCOMES:
correlation between change of CFD value and radiologic response | 2 years
  Confirmation of correlation between CFD change value and imaging response (PR/CR versus SD/PD)
relationship between baseline CFD and tumor marker | 2 years
  Confirmation of relationship between baseline CFD value and other tumor markers (CEA, CA19-9, CA125, PSA) and LDH
correlation between change of CFD value and change of tumor marker | 2 years
  Confirmation of relationship between change of CFD value and change of other tumor markers (CEA, CA19-9, CA125, PSA) and LDH

CONTACTS AND LOCATIONS:
Overall Officials: Kwonoh Park, MD, phD, Principal Investigator — Medical Oncology and Hematology, Department of Internal medicine, Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leon SA, Shapiro B, Sklaroff DM, Yaros MJ. Free DNA in the serum of cancer patients and the effect of therapy. Cancer Res. 1977 Mar;37(3):646-50. PMID 837366
- [Result] Agostini M, Pucciarelli S, Enzo MV, Del Bianco P, Briarava M, Bedin C, Maretto I, Friso ML, Lonardi S, Mescoli C, Toppan P, Urso E, Nitti D. Circulating cell-free DNA: a promising marker of pathologic tumor response in rectal cancer patients receiving preoperative chemoradiotherapy. Ann Surg Oncol. 2011 Sep;18(9):2461-8. doi: 10.1245/s10434-011-1638-y. Epub 2011 Mar 17. PMID 21416156
- [Result] Goldshtein H, Hausmann MJ, Douvdevani A. A rapid direct fluorescent assay for cell-free DNA quantification in biological fluids. Ann Clin Biochem. 2009 Nov;46(Pt 6):488-94. doi: 10.1258/acb.2009.009002. Epub 2009 Sep 3. PMID 19729503
- [Result] Czeiger D, Shaked G, Eini H, Vered I, Belochitski O, Avriel A, Ariad S, Douvdevani A. Measurement of circulating cell-free DNA levels by a new simple fluorescent test in patients with primary colorectal cancer. Am J Clin Pathol. 2011 Feb;135(2):264-70. doi: 10.1309/AJCP4RK2IHVKTTZV. PMID 21228367
- [Result] Kim JJ, Park K, Han YR, Kim SH, Oh SB, Oh SY, Hong YJ, Yun MS. Verification of performance of a direct fluorescent assay for cell-free DNA quantification, stability according to pre-analytical storage conditions, and the effect of freeze-thawing. Biomed Rep. 2021 Aug;15(2):68. doi: 10.3892/br.2021.1444. Epub 2021 Jun 15. PMID 34257964